CLINICAL TRIAL: NCT03517631
Title: A Pilot Study to Evaluate Efficacy and Safety of Multiplexed shRNA-modified CD34+ Cells in HIV-infected Patients.
Brief Title: An Efficacy and Safety Study of shRNA-modified CD34+ Cells in HIV-infected Patients.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: R&D Kanglin Biotech (Other)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL1702
Record Dates: First submitted 2018-03-20; First posted 2018-05-07 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections; AIDS
Keywords: HIV; AIDS; Lentivirus; shRNA; Multiplex; Gene therapy
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Busulfan

STUDY DESIGN:
Intervention Model Description: Infusion of autologous CD34+ cells transduced with shRNAs targeting CCR5 and HIV genome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No busulfan preconditioning (Experimental): shRNA-modified CD34+ cells without busulfan preconditioning.
  Interventions: Biological: shRNA-modified CD34+ cells
- Low dose busulfan preconditioning (Experimental): shRNA-modified CD34+ cells, with a single dose of 1 mg/kg busulfan administered every 6 hours for 4 times as preconditioning for transplantation.
  Interventions: Biological: shRNA-modified CD34+ cells; Drug: Low dose busulfan preconditioning
- High dose busulfan preconditioning (Experimental): shRNA-modified CD34+ cells, with a single dose of 1 mg/kg busulfan administered every 6 hours for 8 times as preconditioning for transplantation.
  Interventions: Biological: shRNA-modified CD34+ cells; Drug: Busulfan preconditioning

INTERVENTIONS:
Biological: shRNA-modified CD34+ cells — Infusion of CD34+ cells transduced with shRNAs.
Drug: Low dose busulfan preconditioning — A single dose of 1 mg/kg busulfan administered every 6 hours for 4 times as preconditioning for transplantation.
  Other Names: Busulfex
  Arms: Low dose busulfan preconditioning
Drug: Busulfan preconditioning — A single dose of 1 mg/kg busulfan administered every 6 hours for 8 times as preconditioning for transplantation.
  Other Names: Busulfex
  Arms: High dose busulfan preconditioning

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of autologous CD34+ cells that stably express multiplexed shRNA to treat HIV infection.

DETAILED DESCRIPTION:
CD34+ cells will be isolated from mobilized PBMC of HIV patients. The cells will be lentivirally transduced with multiplexed shRNAs in the same vector that target CCR5 and HIV genome. Such modified cells will be infused back to the patients who have received bulsufan preconditioning before infusion. The patients will then be evaluated for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) from 18 - 25; body weight ≥50kg.
* Diagnosis of HIV infections/AIDS based on "Diagnostic Criteria for HIV/AIDS" WS 293-2008.
* No antiretroviral therapy (ART) in the past 6 weeks and refuse to receive ART.
* CD4 T cell count ≥350/μl.
* No plan for pregnancy in the near future and agree to practice non-drug based contraception.
* Voluntary to participate in the study, comply with the study design to complete all monitory measurements, and agree to sign the study agreement.

Exclusion Criteria:

* Existence of infections/opportunistic tumors.
* Mutations in the shRNA target sequences.
* White blood cell count <3x10^9/L, neutrophil count <1.5x10^9/L, hemoglobin <110g/L, platelet count <100x10^9/L.
* Liver diseases (HBV, chronic HCV infection, congenital liver metabolic disease), abnormal liver functions (test value 2x above normal).
* Kidney deficiency (Creatinine level above the upper limit of normal levels).
* Severe chronic disease, metabolic disease (e.g., diabetes), neurological and psychiatric diseases.
* History of pancreatitis.
* Women in pregnancy, lactating or at reproductive age who do not practice contraception.
* Allergy to agents or drugs used in the study.
* Verified or suspected abuse of alcohol and drugs.
* Participated in other clinical trials within 3 months.
* Based on investigator's assessment, those who are unfit for the study (e.g., general weakness, poor compliance with study design).
* Personal or family history of tumors.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse side effects | 18 months
  Patients will be monitored for any signs of adverse effects.

SECONDARY OUTCOMES:
Efficacy of treatment | 18 months
  Evaluate the efficacy of modified autologous CD34+ cells by monitoring CD4 counts and HIV-1 RNA level.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Ph.D, Study Director — Caolang Road NO. 2901, Jinshan District, Shanghai
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No